CLINICAL TRIAL: NCT07065461
Title: The Impact of Almond Size in a White Chocolate Matrix on Satiation, Postprandial Glycemia & Lipemia, Chewing Exertion, Eating Rate, and Product Liking: A Randomized Crossover Trial
Brief Title: The Chocolate Almond Study - Relating Chewing to Satiation and Postprandial Response
Acronym: CAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1669; 400819 (Other Grant/Funding Number: Natural Sciences & Engineering Research Council of Canada)
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Satiation, Satiety; Postprandial Glycemia; Postprandial Lipemia
Keywords: Almonds; Particle size; Satiation; Satiety; Postprandial glycemia; Postprandial lipemia; White chocolate; Food matrix; chewing exertion

STUDY DESIGN:
Intervention Model Description: Acute meal postprandial study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Individuals collecting, entering, and analyzing data will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White chocolate with whole almonds (Experimental): Ad libitum serving with 2.25:1 weight per cent chocolate:almonds
  Interventions: Other: 200 g serving of white chocolate-based confection product
- White chocolate without almonds (Experimental): Ad libitum serving
  Interventions: Other: 200 g serving of white chocolate-based confection product
- White chocolate with chopped almonds (Experimental): Ad libitum serving with 2.25:1 weight per cent chocolate:almonds
  Interventions: Other: 200 g serving of white chocolate-based confection product

INTERVENTIONS:
Other: 200 g serving of white chocolate-based confection product — 200 g serving of white chocolate-based confection product

SUMMARY:
The goal of this clinical trial is to relate chewing behaviours to food intake and postprandial response for a texturally complex food matrix (almonds in white chocolate) in healthy young females. The main questions it aims to answer are:

* Does the presence or preparation of almonds (whole versus chopped) influence satiation, i.e., the amount consumed at an ad libitum meal?
* What is the correlation between chewing behaviour, satiation, and changes in postprandial glucose, triacylglycerols, and satiety ratings? Participants will attend the research centre fasted on three occasions to consume an ad libitum meal, complete questionnaires, and provide fasting and postprandial finger prick blood samples.

DETAILED DESCRIPTION:
This study is investigating how the size and presence of almonds (whole vs. chopped) in a white chocolate matrix affect satiation (termination of eating) and postprandial satiety, glycemia, and lipemia. Over three visits, fasted healthy adult female participants will consume three types of white chocolate bark: one with whole almonds, one with chopped almonds, and one with just chocolate. The amount of each ad libitum meal consumed and eating time will be quantified to compare satiation between the confectionery products. Participants will rate their chewing experiences (e.g., exertion, liking, motivations to stop eating) and feelings of satiety up to 180 minutes using paper questionnaires. Participants will also provide finger prick blood samples for determination of glucose and triacylglycerol levels before and after eating each treatment, i.e., at baseline (0 minutes) and 120 (glucose) and 180 (triacylglycerols) minutes after eating. Overall, this study aims to provide insights into the role of food structure in influencing eating and metabolic response and ultimately how food choices can be optimized for better management of blood sugar, satiety, and lipemia to support cardiometabolic health. It is being complemented by a collaboration with researchers in the Department of Food Science at the University of Guelph (led by Prof. Lisa Duizer) examining sensory perception of these same texturally complex foods and the relationship between oral processing behaviour and bolus properties, as well as by in vitro digestion investigations of digestate properties and nutrient release to enable an integrated understanding linking food structure to eating behaviour and postprandial metabolism.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-27.9 kg/m^2 or waist circumference less than 88 cm
* No known food allergies or sensitivities
* Non-restrained eaters based on the Three Factor Eating Questionnaire
* No history of gastrointestinal diseases that may interfere with eating behaviour or digestion
* Not on medications that affect appetite, digestion, blood sugar regulation, saliva production, or chewing
* Stable medication use
* Non-smokers
* Not gained or lost significant weight during the past 3 months
* Regular monthly menstrual cycles
* Not pregnant, lactating, or post-menopausal

Exclusion Criteria:

* Diabetes or other metabolic disorders affecting glycemia and overall cardiometabolic health
* Any food allergies, intolerance, or sensitivities
* Any life-threatening allergy
* Pregnant or breastfeeding
* Participation in another clinical trial
* Alcohol consumption more than 14 drinks per week
* Smokers or those with a smoking history or more than 10 years
* Regular use of recreational drugs (e.g., marijuana, ecstasy, magic mushrooms)
* Restrained eater as defined by > 15 on the Three-Factor Eating Questionnaire
* Unusual sleep patterns
* Irregular breakfast consumption
* Recent weight changes or intended weight loss or gain or having lost or gained >10% of body weight within the last 6 months
* Using medications known to affect appetite, digestion, blood sugar regulation, lipids, or chewing (excluding oral contraceptives)
* Experiences dry mouth, in general or due to medication side effects
* Diagnosed with Sjogren's Syndrome (autoimmune condition linked to severe dry mouth)
* Inability to adhere to study protocols
* Not comfortable providing finger prick blood samples
* Avoids consuming almonds or chocolate
* Has temporomandibular joint disorder (TMJ)
* Has or history or oral cancer
* Recent dental or jaw surgery
* Avoids eating hard foods for concerns of dental fractures or for general oral health
* Individuals with dentures, braces, Invisalign, or other dental implants that cause difficulty chewing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Satiation | Baseline
  Weight (g) of chocolate confection consumed during ad libitum meal

SECONDARY OUTCOMES:
Borg rating of perceived exertion | Immediately after the ad libitum meal is consumed
  Paper scale rating of effort required to chew the meal where 0 = No effort at all and 10 = Very very severe chewing effort
Eating rate | Immediately after the ad libitum meal is consumed
  Calculated from time of eating
Blood glucose | Baseline and 2 hours later
  Based on finger prick blood analysis
Blood triacylglycerols | Baseline and 3 hours later
  Based on finger prick blood analysis
Postprandial satiety visual analogue scale | Baseline until 180 minutes
  Paper questionnaire scale ratings of Hunger, Fullness, Prospective Consumption, and Desire to Eat where each is 100 mm ranging from 0 (minimum) to 100 (maximum). For example, 0 = Not at all Hungry and 100 = As Hungry as Possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Health Sciences, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No